CLINICAL TRIAL: NCT00181831
Title: Proton Magnetic Resonance Spectroscopy in Children and Adolescents With Bipolar Disorder
Brief Title: Spectroscopy in Children and Adolescents With Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Janssen Pharmaceutica (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2002-P-000661
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Disorder; ADHD
Keywords: SPECT; bipolar disorder; ADHD; children
MeSH Terms: conditions — Bipolar Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Proton Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Proton Magnetic Resonance Spectroscopy

SUMMARY:
The primary aim of this study is to use proton magnetic resonance spectroscopy to look at myo-Inositol containing compounds (Ino) and creatine + phosphocreatine (Cr) in the anterior cingulate of 20 children with bipolar disorder between the ages of 6-17 years old free of risperidone treatment and 20 children with bipolar disorder after an eight-week or longer treatment with risperidone. For comparison, results will also be obtained from 20 controls (without bipolar disorder or ADHD) of the same age and gender as well as from 20 children or adolescents with a diagnosis of Attention Deficit Hyperactivity Disorder. We hypothesize that Ino/Cr levels in the anterior cingulate will correlate positively with manic symptoms using the Young mania rating scale (YMRS). Ino/Cr levels in the anterior cingulate in the anterior cingular gyrus will be lower in subjects who have received eight weeks or longer of risperidone

DETAILED DESCRIPTION:
Choline containing compound (Cho) and creatine + phosphocreatine (Cr) have been found to be greater in the orbitofrontal cortex of depressed adolescents. In addition, Cho/Cr has been found to increase in the anterior cingulate in depressed patients with bipolar affective disorder (BPD) compared with comparison subjects. Also, BPD subjects not taking antidepressants had a significantly higher anterior cingulate Cho/Cr compared with subjects taking antidepressants or comparison subjects. Therefore it would appear the frontal lobe Cho/Cr is increased in depression. Given these findings, we are interested in looking at subjects with mania to investigate if there may also be a biological marker for mania and drug response. Mania measured using the YMRS have been associated with an increase in the anterior cingulate Ino/Cr in manic children, adolescents, and adults with bipolar affective disorder. In addition, children and adolescents who were responsive to lithium showed a decrease in Ino/Cr levels after acute lithium treatment. We will test whether Ino/Cr levels will correlate positively with manic symptoms using the YMRS, as well as whether overall Ino/Cr levels will be lower for children and adolescents receiving risperidone.

The primary aim of this study is to use proton magnetic resonance spectroscopy to look at myo-Inositol containing compounds (Ino) and creatine + phosphocreatine (Cr) in the anterior cingulate of 20 children with bipolar disorder between the ages of 6-17 years old free of risperidone treatment and 20 children with bipolar disorder after an eight-week or longer treatment with risperidone. For comparison, results will also be obtained from 20 controls (without bipolar disorder or ADHD) of the same age and gender as well as from 20 children or adolescents with a diagnosis of Attention Deficit Hyperactivity Disorder. We hypothesize that Ino/Cr levels in the anterior cingulate will correlate positively with manic symptoms using the Young mania rating scale (YMRS). Ino/Cr levels in the anterior cingulate in the anterior cingular gyrus will be lower in subjects who have received eight weeks or longer of risperidone

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 6-17 years of age
2. Subject and parent must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol
3. Subjects and their legal representatives must be considered reliable
4. Each subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document.
5. Bipolar subjects must have a diagnosis of bipolar I or bipolar II disorder with a lifetime manic or mixed episode (with or without psychotic features) according to the DSM-IV confirmed by structured diagnostic interview (KSADS)
6. ADHD subjects must meet full criteria for ADHD (with or without hyperactivity) according to the DSM-IV confirmed by structured diagnostic interview (KSADS)

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Pregnant of nursing females
3. Presence of metal or surgical devices (aneurysm clips, metal plates, cochlear implants, neurostimulators, braces, and other items) in vital areas.
4. Severe phobia of being in small, enclosed spaces (claustrophobic)
5. Bipolar subjects must either have been free of antipsychotic medication (including risperidone) for 3 months of longer OR be currently treated with risperidone for 8 weeks or longer.
6. ADHD subjects must not meet criteria for bipolar disorder by structured interview (KSADS). These subjects must be free of antipsychotic medication for 3 months or longer).
7. Control subjects must not meet criteria for ADHD or bipolar disorder by structured interview (KSADS). These subjects must be free of antipsychotic medication treatment for 3 months or longer.
8. Left hand dominant subjects will be excluded

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 20 children with bipolar disorder between the ages of 6-17 years old free of risperidone treatment and 20 children with bipolar disorder after an eight-week or longer treatment with risperidone.
Sampling Method: Non-Probability Sample
Enrollment: 80
Dates: Start 2002-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States